CLINICAL TRIAL: NCT05888558
Title: Screening of Serum Exosomal miRNA as a Biomarker for Ocular Muscle Myasthenia
Brief Title: Screening of Serum Exosomal miRNA as a Biomarker for Ocular Muscle Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, XiaoYong Liu, Doctor, First Affiliated Hospital of Jinan University
Other Study IDs: 2021.11JinanU
Record Dates: First submitted 2021-11-04; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Myasthenia Gravis
Keywords: Ocular myasthenia gravis;; miRNA; exosomes
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ocular myasthenia gravis group: Ocular myasthenia gravis,age between 18-50 years old
  Interventions: Device: Body fluid diagnosis
- General myasthenia gravis group: General myasthenia gravis,age between 18-50 years old
  Interventions: Device: Body fluid diagnosis
- Healthy control group: people who are healthy without any systemic diseases，18-50 years old
  Interventions: Device: Body fluid diagnosis

INTERVENTIONS:
Device: Body fluid diagnosis — miRNAs derived from exosomes in the serum

SUMMARY:
Ocular muscle myasthenia gravis (Ocular Myasthenia Gravis, OMG) has a high incidence and is difficult to diagnose. It is very necessary to find specific diagnostic indicators for OMG. By collecting peripheral blood of OMG, systemic myasthenia gravis and healthy people, extract miRNAs derived from exosomes in the serum and perform high-throughput sequencing, then use bioinformatics analysis methods to screen specifically expressed miRNAs as biomarkers for OMG diagnosis .

DETAILED DESCRIPTION:
Part I: (1) Collect peripheral blood samples from patients with early-onset OMG, early-onset GMG and healthy subjects of age and sex matched who have been diagnosed for the first time and have not undergone any drug treatment. There are 6 cases in each group. Extract the secretion miRNA in serum and conduct high-throughput sequencing. Analyze and compare the differential expression miRNAs between OMG, GMG and healthy control groups by edgeR. The standard of differential expression is set as | logFC |>1, p<0.05. Use miRTarBase, TargetScan, and miRDB to predict target genes for differentially expressed miRNAs. Conduct GO enrichment and KEGG signaling pathway analysis on target genes. The STRING tool is used to construct the target gene protein interaction network (PPI). According to the importance of the target gene calculated by the maximum population concentration ratio (MCC) method, the top ten genes (hub genes) are selected and analyzed.

(2) Randomly collect peripheral blood samples from patients with early-onset OMG, early-onset GMG, and age-matched healthy subjects, with 10 samples in each group. The differentially expressed miRNAs obtained during the sequencing phase were validated using real-time fluorescence quantification (RT-qPCR). Construct a receiver operating characteristic curve (ROC) curve to evaluate the diagnostic efficacy of the identified miRNA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical manifestations: fluctuating myasthenia;

  * neostigmine test positive; ③ AChR-Ab, Musk-Ab, LRP4-Ab antibodies positive; ④repetitive nerve stimulation or single fiber EMG Positive (comply with the first one of the above diagnostic criteria and any one of the other three, and at the same time exclude ophthalmoplegia caused by other diseases, the diagnosis can be confirmed).

Exclusion Criteria:

①Combined with other autoimmune diseases or other inflammatory diseases; ②Patients with tumorous diseases;

* Received targeted biologics, intravenous gamma globulin, plasma exchange therapy within three months before treatment; ④Pregnancy Status or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People within age 18-50 years old who is diagnosed with OMG,GMG or healthy people.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-07-04 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
A specific miRNA maybe miR-340-5p，miR-106b-5p or miR-27a-3p is a biological marker for diagnosis of OMG | 12,2022
  find some specific miRNA to diagnose OMG.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes